CLINICAL TRIAL: NCT02094794
Title: Phase II Study of Total Marrow and Lymphoid Irradiation (TMLI) Given in Combination With Cyclophosphamide and Etoposide as Conditioning for Allogeneic (HSCT) in Patients With High-Risk Acute Lymphocytic or Myelogenous Leukemia
Brief Title: Total Marrow and Lymphoid Irradiation and Chemotherapy Before DSCT in Treating Patients With High-Risk ALL or AML
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14012; NCI-2014-00639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14012 (Other: City of Hope Medical Center); R01CA154491 (NIH)
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Etoposide; Cyclophosphamide; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (TMLI, chemotherapy) (Experimental): Patients undergo image guided TMLI on days -9 to -5, receive etoposide IV on day -4 and cyclophosphamide IV on day -2, and undergo allogeneic peripheral blood stem cell or bone marrow transplant on day 0.
  Interventions: Drug: etoposide; Drug: cyclophosphamide; Radiation: total marrow irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: allogeneic bone marrow transplantation

INTERVENTIONS:
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Radiation: total marrow irradiation — Undergo TMLI
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic peripheral blood stem cell or bone marrow transplant
Procedure: allogeneic bone marrow transplantation — Undergo allogeneic peripheral blood stem cell or bone marrow transplant
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow

SUMMARY:
This phase II trial studies the safety and efficacy of total marrow and lymphoid irradiation (TMLI) in combination with two chemotherapy drugs, etoposide and cyclophosphamide, as a preparative regimen before donor stem cell transplant in treating patients with high-risk acute lymphocytic leukemia (ALL) or acute myeloid leukemia (AML) who have failed previous therapy. Intensity-modulated radiation therapy (IMRT) uses imaging to provide a three-dimensional view of the area to be irradiated. Doctors can then shape and direct the radiation beams at the area from multiple directions while avoiding, as much as possible, nearby organs. TMLI is a method of using IMRT to direct radiation to the bone marrow. Radiation therapy is given before transplant to suppress the immune system, prevent rejection of the transplanted cells, and wipe out any remaining cancer cells. TMLI may allow a greater radiation dose to be delivered to the bone marrow as a preparative regimen before transplant while causing fewer side effects than standard radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Following a patient safety lead-in, evaluate the anti-tumor activity of the allogeneic hematopoietic cell transplant (alloHCT) preparative regimen - TMLI, cyclophosphamide (Cy) and etoposide (VP-16), as assessed by 2-year progression-free survival (PFS).

SECONDARY OBJECTIVES: I. Estimate overall survival (OS), cumulative incidence (CI) of relapse/progression, and non-relapse mortality (NRM) at 100 days, 1 year and 2 years.

II. Evaluate early and late toxicities/complications by organ and severity, and characterize by organ dose/dose volume, including acute/chronic graft-versus-host-disease (GVHD), infection, and longer-term complications (via protocol #s 07173 and 00029).

OUTLINE: Patients undergo image guided TMLI on days -9 to -5, receive etoposide intravenously (IV) on day -4 and cyclophosphamide IV on day -2, and undergo allogeneic peripheral blood stem cell or bone marrow transplant on day 0.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant has the ability and the willingness to sign the informed consent document (for adults only, for participants with mild cognitive abilities may use a legally authorized representative)
* Documented (signed) informed consent; the patient, family member and transplant staff physician (physician, nurse, and social worker) meet at least once prior to starting the transplant procedure; during this meeting all pertinent information with respect to risks and benefits to donor and recipient will be presented; alternative treatment modalities will be discussed; the risks are explained in detail in the enclosed consent forms
* Karnofsky performance status >= 70% =< 2
* Acute lymphocytic leukemia or acute myelogenous leukemia who are not in first remission or second remission i.e. after failing induction therapy, or in relapse or beyond second remission; (prior therapy with VP-16 and Cytoxan is allowed)
* All candidates for this study must have a human leukocyte antigen (HLA) (A, B, C, DR) identical siblings who is willing to donate bone marrow or primed blood stem cells or a 10/10 allele matched unrelated donor; a single allele mismatch at A, B, C, DR or DQ and a killer immunoglobulin-like receptor (KIR) mismatch at C will be allowed; all ABO blood group combinations of the donor/recipient are acceptable
* The time from the end last induction, re-induction, or consolidation regimen should be greater than or equal to 14 days from planned start of study treatment; Note: Chemotherapy given within 14 days of planned study enrollment for the purpose of controlling counts is permitted
* Total bilirubin =< 1.5 x upper limit of normal (ULN) OR 3 x ULN for Gilbert's disease
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 5 x ULN
* Measured creatinine clearance >= 80 ml/min per 24 hour urine collection OR serum creatinine =< 1.3 mg/dL
* Women of child bearing potential only: Negative urine or serum pregnancy test
* Pulmonary function tests: Forced expiratory volume in one second (FEV1) and carbon monoxide diffusion capacity (DLCO) (adjusted for Hb) >= 50% adjusted of predicted normal value
* Echocardiogram (ECHO) or multi gated acquisition scan (MUGA): ejection fraction of >= 50% AND no finding of abnormal wall motion (i.e. report does not indicate that wall motion is "abnormal" or "altered")
* Electrocardiogram (EKG) showing no ischemic changes and no abnormal rhythm
* Agreement of men AND women-of-child-bearing-potential to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* DONOR ELIGIBILITY: Donor evaluation and eligibility will be assessed as per current City of Hope standard operating procedure (SOP)

Exclusion Criteria:

* Prior autologous or allogeneic hematopoietic stem cell
* Prior radiation therapy that would exclude the use of TMLI
* Plans during the trial to receive any other (non-trial) investigational agents, or concurrent biological, chemotherapy, or radiation therapy; (chemotherapy for white blood count control is permitted)
* Uncontrolled illness including ongoing or active infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to etoposide
* Patients with other active malignancies are ineligible for this study, other than localized malignancies
* Patients with psychological or medical condition that patient's physician deems unacceptable to proceed to allogeneic hematopoietic stem cell transplantation
* Women who are planning to become pregnant or breast feed during the trial
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity, scored on both the Bearman Scale and National Cancer Institute Common Terminology Criteria version 4.03 (Safety lead-in segment) | Up to 30 days after stem cell infusion
  Toxicity information recorded will include the type, severity, and the probable association with the study regimen.
PFS | The time from start of protocol therapy to death, relapse/progression, or last follow-up, whichever comes first, assessed up to 2 years
  Calculated using the Kaplan-Meier method. The cumulative incidence of relapse/progression will be calculated as a competing risk using the Gray method.

SECONDARY OUTCOMES:
OS | The time from start of protocol therapy to death, or last follow-up, whichever comes first, assessed up to 5 years
  Calculated using the Kaplan-Meier method.
Time to relapse/progression | From start of therapy to time of relapse/progression, assessed up to 5 years
  Calculated using the Kaplan-Meier method.
Complete response (CR) proportion | The start of therapy to the time of CR, assessed at day 30
NRM | From start of therapy until non-disease related death, or last follow-up, whichever comes first, assessed up to 5 years
  Calculated using the Kaplan-Meier method. The cumulative incidence of non-relapse mortality will be calculated as a competing risk using the Gray method.
Incidence of infection | Up to 100 days post-transplant
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any.
Incidence of toxicities, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to day 100 post-transplant
  The worst grade of all toxicities will be collected from day -9 to day -1 and again from day 0 to day 30 post-transplant. From day 31 to 100 post-transplant only grade 3, 4 and 5 toxicities will be collected. Toxicity information recorded will include the type, severity, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity. Baseline information (e.g. the extent of prior therapy) and demographic information will be presented.
Incidence of acute graft versus host disease GVHD (aGVHD) of grades 2-4, graded according to the Consensus Grading | Up to day 100 post-transplant
  The first day of acute GVHD onset at a certain grade will be used to calculate cumulative incidence curves for that GVHD grade.
Incidence of aGVHD of grades 3-4, graded according to the Consensus Grading | Up to day 100 post-transplant
  The first day of acute GVHD onset at a certain grade will be used to calculate cumulative incidence curves for that GVHD grade.
Incidence of chronic GVHD, scored according to National Institute of Health Consensus staging | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Stein, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States